CLINICAL TRIAL: NCT07198581
Title: A Randomized Controlled Trial of AI-Assisted Chemotherapy Side Effect Management in Solid Tumor Patients
Brief Title: AI-Assisted Chemotherapy Side Effect Management
Acronym: ALLIANCE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Incheon St.Mary's Hospital (Other)
Responsible Party: Principal Investigator, Young-Joon Kang, Assistant Professor, Incheon St.Mary's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ALLIANCE
Record Dates: First submitted 2025-09-03; First posted 2025-09-30 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer; Colorectal Cancer
Keywords: Large Language Model; LLM; Breast cancer; Side effect; Supportive care; colorectal cancer
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LLM Intervention Group (Experimental): Patients receive standard chemotherapy with AI-assisted symptom management. Healthcare providers input anonymized patient symptoms into a large language model system during clinic visits. The LLM generates management recommendations that physicians review and consider for treatment decisions.
  Interventions: Behavioral: LLM-assisted chemotherapy side effect management
- Standard Care Group (No Intervention): Patients receive standard chemotherapy with conventional symptom management based on institutional protocols and physician clinical judgment.

INTERVENTIONS:
Behavioral: LLM-assisted chemotherapy side effect management — Healthcare providers collect patient symptoms during clinic visits, anonymize the information, and input it into the LLM system via temporary chat sessions. The LLM generates management recommendations which physicians review and consider when adjusting treatment plans. Healthcare providers anonymize patient information and input into LLM using temporary chat sessions. LLM recommendations serve as reference only, with physicians making all final clinical decisions.
  Arms: LLM Intervention Group

SUMMARY:
This two-stage adaptive randomized controlled trial evaluates the feasibility and preliminary efficacy of large language model (LLM)-assisted intervention for managing chemotherapy side effects in patients with solid tumors. Adults with histologically confirmed breast or colorectal cancer scheduled for at least 3 months of systemic chemotherapy will be randomly assigned (1:1) to receive either LLM-assisted care or standard care.

The study employs an adaptive design with initial enrollment of 40 patients (20 per arm), followed by interim analysis. If predefined criteria are met, an additional 134 patients will be enrolled for a maximum total of 174 patients (87 per arm).

In the intervention group, healthcare providers input anonymized patient symptom data into an LLM system using sessions where data is not retained, which generates evidence-based management recommendations. Physicians critically review these recommendations and use them as reference for clinical decision-making, with final treatment decisions remaining under physician discretion. The control group receives standard supportive care without LLM assistance.

The primary outcome is change in health-related quality of life measured by EORTC QLQ-C30 global health status/QoL scale from baseline to end of treatment. Secondary outcomes include proportion achieving clinically meaningful improvement (≥8-point increase), treatment adherence, dose intensity, healthcare resource utilization, and physician acceptance of LLM recommendations.

DETAILED DESCRIPTION:
Chemotherapy-induced side effects affect patient quality of life and treatment outcomes. Studies indicate 86% of patients receiving chemotherapy experience at least one side effect, with 30% reporting moderate to severe symptoms. Common adverse effects including nausea, vomiting, fatigue, anorexia, pain, diarrhea, constipation, mucositis, and peripheral neuropathy lead to dose reductions, treatment delays, or discontinuation.

Care gaps persist despite advances in supportive care due to clinician time constraints and variable attention to specific side effects. Digital health interventions have demonstrated improved quality of life, reduced emergency department visits, and enhanced survival in cancer patients. A 2025 umbrella review reported positive effects of digital health interventions on multiple mental health indicators in cancer patients.

LLMs offer natural language processing and medical knowledge bases. Clinical application remains limited, with only 5% of LLM healthcare studies involving actual patient care according to recent systematic reviews. Reliability concerns and hallucination require physician oversight. While healthcare providers manage life-threatening chemotherapy toxicities effectively, less attention may be given to symptoms that impact quality of life without immediate life-threatening consequences.

This adaptive randomized controlled trial employs a two-stage design. Stage 1 enrolls 40 patients (20 per arm) with breast or colorectal cancer without malignancy-related symptoms at baseline. Stratification occurs by cancer type. The intervention involves healthcare providers collecting patient symptoms during clinic visits, excluding information that could identify patients, anonymizing information according to standardized prompts, and inputting data into the LLM system via temporary chat sessions where no records are retained. The LLM generates symptom analysis and management recommendations. Physicians review recommendations and adjust treatment plans accordingly, with all final decisions remaining under physician responsibility.

Interim analysis after 40 patients are enrolled evaluates safety, feasibility, and efficacy. Safety assessment includes stopping for serious LLM-related issues. Feasibility assessment examines LLM system usage rate (<60% triggers system improvement or additional training) and physician satisfaction. Efficacy assessment evaluates observed effect size and variability, considering study discontinuation only if control group clearly superior or serious harm observed. Based on interim results, up to 134 additional patients may be enrolled for a maximum total of 174 participants.

The primary analysis uses linear mixed-effects models adjusting for baseline scores and stratification factors. A clinically meaningful difference of 8 points on the EORTC QLQ-C30 scale with standard deviation of 20 points provides >85% power at the final sample size. Secondary analyses include logistic regression for clinically meaningful improvement rates, appropriate statistical tests for adherence and toxicity outcomes, and Poisson/negative binomial regression for healthcare utilization.

This study aims to evaluate whether LLM-assisted intervention improves patient outcomes and healthcare resource utilization in oncology practice, providing evidence for the clinical application of LLMs as decision support tools in patient care.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years old) diagnosed with histologically confirmed solid malignancies (breast cancer, colorectal cancer)
* Patients scheduled to receive at least 3 months of systemic chemotherapy
* ECOG performance status 0-2

Exclusion Criteria:

* Severe psychiatric disorders
* Cognitive impairment affecting ability to report symptoms
* Presence of cancer-related symptoms prior to chemotherapy initiation
* Concurrent participation in trials evaluating other symptom management interventions Inability to provide informed consent Life expectancy less than 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2025-11-12 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Change in health-related quality of life measured by EORTC QLQ-C30 global health status/QoL scale (European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 - Global Health Status/Quality of Life Scale) | Baseline, mid-treatment, end of treatment, 3 months post-treatment (up to 9 months)
  Change in health-related quality of life measured by EORTC QLQ-C30 global health status/QoL scale (range 0-100, higher scores indicate better outcomes; less decline indicates better outcomes)

SECONDARY OUTCOMES:
Proportion of patients with ≥8 points improvement in EORTC QLQ-C30 global health status/QoL scale | Baseline, mid-treatment, end of treatment, 3 months post-treatment (up to 9 months)
Proportion of patients completing all planned chemotherapy cycles | Throughout chemotherapy treatment period (approximately 3-6 months)
Relative dose intensity (percentage of planned dose actually administered) | Throughout chemotherapy treatment period (approximately 3-6 months)
Frequency of grade 3-4 toxicities according to CTCAE v5.0 | Throughout chemotherapy treatment period (approximately 3-6 months)
Number of emergency department visits and unplanned hospitalizations | From baseline through 3 months after treatment completion (up to 9 months)
Physician survey with LLM recommendations (intervention arm only) | Monthly during treatment and at end of treatment, up to 6 months
  Mean physician usefulness score for LLM recommendations assessed by physician evaluation survey (1-5 point scale) (intervention arm only)

CONTACTS AND LOCATIONS:
Locations (1):
- Incheon St. Mary's Hospital, College of Medicine, The Catholic University of Korea, Incheon, South Korea